CLINICAL TRIAL: NCT05234138
Title: Generation Of a Lung Biobank for Future Use
Acronym: GOLF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4977
Record Dates: First submitted 2020-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA and Streck (40ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Sample — Blood Sample

SUMMARY:
The aim is to invite 1,000 patients with symptoms triggering the lung cancer diagnostic pathway or with significant risks of lung cancer, referred to The Royal Marsden NHS Foundation Trust (RMH) referral centres (Kingston Hospital NHS Foundation Trust, Epsom and St Helier University Hospitals NHS Trust, Croydon University Hospitals NHS Foundation Trust or St George's University Hospitals NHS Foundation Trust) over a 1 year period, to complete a life style questionnaire, document lung function tests and to donate a blood sample for storage with a view to testing for a genetic signature and other biomarkers in future studies from this established biobank.

DETAILED DESCRIPTION:
Patients will have been referred under the two week rule (TWR) diagnostic pathway, some will have lung cancer, others not, and other patients will have had a diagnosis of lung cancer by other pathways i.e. non TWR.

There are 3 groups of patients:

Group A - lung cancer patients at any stage and by any non TWR pathway, n=250. Group B - lung cancer patients who were referred initially by the TWR pathway, n=150.

Group C - Subjects referred by the TWR pathway (i.e. with symptoms) who do not have lung cancer, or subjects referred by any pathway who do not have lung cancer but do have radiological changes (that need follow up) or a strong family history of lung cancer, n=600.

A strong family history for this study means 1 or more first degree relatives with lung cancer with at least one individual having lung cancer at age <50 yrs.

ELIGIBILITY:
Inclusion Criteria:

One of the following criteria:

* Patients with lung cancer at any stage or time in their disease.
* Patients without lung cancer who have been referred by the TWR pathway.
* Patients without lung cancer who have radiological changes on their X-Ray or CT scan that need follow up.
* Patients without lung cancer who have a strong family history of lung cancer. PLUS
* Patients aged >18 Years
* Patients who have signed informed consent form

Exclusion Criteria:

* Unable to provide informed consent.
* Bleeding disorder or other medical condition that would make a blood sample hazardous.
* Within 3 weeks of chemotherapy or radiotherapy (as low lymphocyte may be associated with poor DNA yield).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Royal Marsden Hospital NHS Foundation Trust (Sutton and Chelsea)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Create a collection of blood samples in a Biobank for Future Use | 3 Years
  The aim is to ask 1,000 patients with symptoms triggering the lung cancer diagnostic pathway or with significant risks of lung cancer and to create a collection of blood samples in a Biobank for Future Use.
Feasibility as a Primary Endpoint | 3 Years
  Feasibility will be reported as the primary endpoint, where we expect 50% of patients would be willing to give a blood sample- i.e. 250/year for 2 years and thus a biobank will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom